CLINICAL TRIAL: NCT04966208
Title: Root Coverage Using Tunneling Technique of Xenogenic Collagen Matrix vs. Autologous Connective Tissue as a Treatment of Miller Class Two Gingival Recession (RCT Study)
Brief Title: Gingival Recession Treatment Using Two Different Surgical Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mortada, Lecturer of Periodontology and Oral Implantology-Faculty of Dentistry, Assiut University, Egypt., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDBSUREC/08042021/FA
Record Dates: First submitted 2021-06-21; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Gingival Recession; Root Planing
Keywords: root coverage; mucoderm; connective tissue; grafts
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- root coverage surgeries using autologous connective tissue for treatment of gingival recession (Active Comparator): root coverage surgeries using tunneling technique of autologous connective tissue as a treatment of Miller class two gingival recession
  Interventions: Procedure: xenogeneic collagen matrix
- root coverage surgeries using xenogenic collagen matrix for treatment of gingival recession (Experimental): root coverage surgeries using tunneling technique of mucodrm membrane ; xenogeneic collagen matrix as a treatment of Miller class two gingival recession
  Interventions: Procedure: xenogeneic collagen matrix

INTERVENTIONS:
Procedure: xenogeneic collagen matrix — xenogeneic collagen matrix called mucoderm used for root coverage for treatment of gingival recession instead of harvesting from the patients connective tissue

SUMMARY:
Coronally the advanced flap is considered a predictable treatment of gingival recession but in certain situations, it needs a filler like subperiosteal connective tissue graft (CTG) which is considered as the gold standard treatment approach.

This randomized controlled trial compares the clinical benefits and effectiveness of a xenogenic collagen matrix (mucoderm, botiss, dental, Berlin, Germany) as a filler to the subperiosteal connective tissue graft (CTG).

ELIGIBILITY:
Inclusion Criteria:

* -The selected patients for this study are non-smokers, aged 18-60 years with multiple gingival recession (Miller class 1, or 2.) for more than two adjacent affected teeth with plaque score less than 25%

Exclusion Criteria:

* -Patients with systemic complications, psychological problems, parafunctional habits, or patients presented with Mal-posed teeth, hypermobile teeth, teeth with Miller class 3 gingival recession were excluded from this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
The zone of keratinized gingiva | 6 months after the surgery
  The distance from the tip of the papilla to the mucogingival junction minus the probing depth measured in mm using graduated periodontal probe.

SECONDARY OUTCOMES:
Periodontal probing depth | 6 months after the surgery
  measured from the gingival margin to the depth of the gingival sulcus in six sites per tooth and measured in mm.
Clinical attachment loss | 6 months after the surgery
  measured from the cementoenamel junction to the depth of the sulcus in six sites per tooth and measured in mm.
Gingival recession | 6 months after the surgery
  The depth measured from the gingival margin to the cementoenamel junction in mm.
Patient satisfaction of the esthetics | 6 months
  measured using the visual analog scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No